CLINICAL TRIAL: NCT05471102
Title: Role of Ligation of the Anterior Division of the Internal Iliac Artery in Conservative Management of Patients Diagnosed With Partial or Focal Placenta Accreta Spectrum
Brief Title: Ligation of Anterior Internal Iliac Artery With Conservative Management of Partial or Focal Placenta Accreta Spectrum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdalla Mousa, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS-38-2022
Record Dates: First submitted 2022-07-03; First posted 2022-07-22 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator): Cases managed by uterine lower segment resection with ligation ((suturing)) of the anterior division of the internal iliac artery (4 cm distal to the bifurcation of the common iliac artery); in addition to the bilateral uterine artery ligation at 2 levels; bilateral ligation at a level below the lower most placental part followed by bilateral uterine artery ligation at the level of the hysterotomy incision.
  Interventions: Procedure: Study group: lower segment resection with ligation of the anterior division of the internal iliac artery
- Control group (Placebo Comparator): Cases managed by uterine lower segment resection without ligation of the anterior division of the internal iliac artery. (i.e., only bilateral ligation at a level below the lower most placental part followed by bilateral uterine artery ligation at the level of the hysterotomy incision).
  Interventions: Procedure: Control group: lower segment resection without ligation of the anterior division of the internal iliac artery

INTERVENTIONS:
Procedure: Study group: lower segment resection with ligation of the anterior division of the internal iliac artery — Cases managed by uterine lower segment resection with ligation ((suturing)) of the anterior division of the internal iliac artery (4 cm distal to the bifurcation of the common iliac artery); in addition to the bilateral uterine artery ligation at 2 levels; bilateral ligation at a level below the lower most placental part followed by bilateral uterine artery ligation at the level of the hysterotomy incision.
  Arms: Study group
Procedure: Control group: lower segment resection without ligation of the anterior division of the internal iliac artery — Cases managed by uterine lower segment resection without ligation of the anterior division of the internal iliac artery. (i.e., only bilateral ligation at a level below the lower most placental part followed by bilateral uterine artery ligation at the level of the hysterotomy incision).
  Arms: Control group

SUMMARY:
The patients will be divided into 2 groups:

Group (A) - Study group: Cases managed by lower segment resection with ligation of the anterior division of the internal iliac artery

Group (B) - Control group: Cases managed by lower segment resection without ligation of the anterior division of the internal iliac artery

The following operative details will be recorded:

* Estimation of total blood loss
* Pre and 24-h post-operative hemoglobin (g/dl).
* The need for blood transfusion and its amount intra or postoperative will be recorded
* Operative time and postoperative hospital stay will be recorded.
* Close post-operative monitoring of the patients' vital signs, drain output, and urine output
* Presence or absence of intraoperative complications; bladder, ureteric, bowel, or vascular injuries will be recorded.
* Monitoring for postoperative morbidities

DETAILED DESCRIPTION:
The patients will be divided into 2 groups:

Group (A) - Study group: Cases managed by uterine lower segment resection with ligation of the anterior division of the internal iliac artery (4 cm distal to the bifurcation of the common iliac artery).

Group (B) - Control group: Cases managed by uterine lower segment resection without ligation of the anterior division of the internal iliac artery.

In both groups, bilateral uterine artery ligation at 2 levels will be done; bilateral ligation at a level below the lower most placental part, followed by bilateral uterine artery ligation at the level of the hysterotomy incision.

The following operative details will be recorded:

* Estimation of total blood loss
* Pre and 24-h post-operative hemoglobin (g/dl).
* The need for blood transfusion and its amount intra or post-operative will be recorded
* Operative time and postoperative hospital stay will be recorded.
* Close post-operative monitoring of the patients' vital signs, drain output, and urine output
* Presence or absence of intraoperative complications; bladder, ureteric, bowel, or vascular injuries will be recorded.
* Monitoring for postoperative morbidities

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-40 years old.
* Pregnancy of singleton living fetus.
* Previous one or more cesarean sections.
* Gestational age: > 36 weeks.
* Elective termination of pregnancy.
* Cases not requiring preoperative blood transfusion.
* Cases with focal area of placental adherence or invasion leaving sufficient healthy myometrial tissue for uterine repair and preservation.
* The following ultrasound markers such as "loss of clear retroplacental translucency", "myometrial thinning", "abnormal lacunae", "irregular bladder wall", "utero-vesical hypervascularity".

Exclusion Criteria:

* Multifetal pregnancy.
* More than four previous sections.
* Emergency termination of pregnancy due to antepartum hemorrhage, placental separation or rupture uterus.
* Intrauterine fetal death.
* Women with history of any medical disorder with pregnancy eg. Gestational diabetes and hypertension.
* Premature rupture of membranes.
* Cases misdiagnosed as placenta accreta by ultrasound preoperatively, and spontaneous full placental separation occurred intraoperative. "will be excluded before randomization"
* Cases with PAS with total invasion involving all placental lobules.
* Cases who will be managed by cesarean hysterectomy due to uncontrolled intraoperative bleeding.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2022-07-03 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Amount of blood loss intra-operative | during operation
  Amount of blood loss intra-operative
Amount of blood loss 24 hours post-operative | 24 hours post-operative
  Amount of blood loss 24 hours post-operative

SECONDARY OUTCOMES:
Operative time | during operation
  duration of the surgery
Number of blood units transfused | within 24 hours after surgery
  Number of blood units transfused within 24 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt